CLINICAL TRIAL: NCT04764396
Title: Assessing Effects of Heparin Priming and Pass Number on Tissue Quality of Fine Needle Biopsies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding and change in research direction.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jorge Machicado, MD, MPH, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00172203
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Pancreas; Mass Lesion
Keywords: biopsy; pancreas lesion; endoscopic fine needle biopsy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: After the amendment (Ame00126774) 98 more participants will be randomized.
Who Masked: Participant, Outcomes Assessor
Masking Description: The pathologist will be blinded to the allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Heparin priming biopsies (Experimental)
  Interventions: Combination Product: Heparin will be used for needle priming (BD PosiFlush™ Pre-Filled Heparin Lock Flush Syringe)
- Standard of care (saline) (Active Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Combination Product: Heparin will be used for needle priming (BD PosiFlush™ Pre-Filled Heparin Lock Flush Syringe) — The fine needle biopsy (FNB) needle will be flushed with 1 mL of heparin (100 USP/mL) and then flushed with air. Pass 1, 2, and 3 will be collected in separate jars and sent to pathology, as per standard clinical procedures. Between passes, after tissue is extracted from the needle, the needle will be flushed with 1 mL of heparin (100 USP/mL) and flushed with air before next pass is made.
  Arms: Heparin priming biopsies
Drug: Saline — FNB will be performed as current standard methods in the medical procedure unit without the use of heparin priming. Pass 1, 2, and 3 will be collected in separate jars and sent to pathology, as per standard clinical procedures. Between passes, after tissue is extracted from the needle, the needle will be flushed saline and or air as per current standards of care.
  Arms: Standard of care (saline)

SUMMARY:
This is a randomized study that will enroll patients scheduled for an endoscopic ultrasound biopsy of a pancreas lesion to be in the heparin or saline group during the procedure.

The purpose of this study is to examine the effect of blood contamination, heparin priming of the fine needle biopsies, and pass number on tumor tissue quality in fine needle biopsies.

The hypothesis for this study is that fine needle biopsy tissue quality of pancreatic masses decreases with increasing pass number due to blood contamination; this blood contamination can be ameliorated with priming of the needle with an anticoagulant such as heparin.

DETAILED DESCRIPTION:
A total of 3 fine-needle biopsy passes will be performed on every procedure. The tissue specimens from each of the 3 passes will be collected in 3 separate jars of 10% formalin for tissue analysis. The use of heparin flushing vs. not heparin flushing will be based on their randomized group assignments.

In the heparin arm, between passes, after tissue is extracted from the needle, the needle will be flushed with 1 mL of heparin (100 USP/mL) and flushed with air before the next pass will be made. This means the needle will have no heparin during the first pass. In the standard of care arm, between passes, after tissue is extracted from the needle, the needle will be flushed with saline and/or air as per current standards of care.

This study was amended at the Institutional Review Board (IRB) after having enrolled only two participants. Following the amendment, the responsible party changed and with that change some adjustments were made to the interventions, analysis and some outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient identified as having a possible solid pancreatic lesion on computed tomography or magnetic resonance
* Patient scheduled for Endoscopic ultrasound (EUS) for sampling of pancreatic mass

Exclusion Criteria:

* known history of coagulopathy
* history of heparin allergy
* patients with evidence of vascular tumors on imaging
* Patients with history of chronic pancreatitis
* Pregnant patients
* Medically unstable patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2021-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Machicado, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) and related data dictionaries available. All IPD that underlie results in our planned publication, after deidentification. IPD will be uploaded to a data repository to be determined at time of publication.
Supporting Information: Study Protocol, SAP
Time Frame: IPD will be available beginning 3 months following article publication and at a minimal ending 5 years following article publication.
Access Criteria: Anyone who wishes to access the data may do so, following the requirements specified by the repository.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Started | 1 | 1
Completed | 0 | 1
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline) | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Customized [Count of Participants; unit: Participants]
  Age 18 - 85 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 0 | 1 | 1
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cellularity Captured in Fine Needle Biopsies for the Heparin Group
Description: Hematoxylin and eosin (H&E) slides from the passes 1, 2, and 3 will be compared. The number of cells present on each H&E slide will be quantified by using image processing software. This value will be total number of cells divided by the total area of the biopsy.
Time Frame: Day 1 (biopsy tissue obtained)
Population: No data is presented here because, with only 1 participant per arm, it is impossible to share this data, as doing so would conflict with the required informed consent language for ACTs, which says, "This website [ClinicalTrials.gov] will not include information that can identify you" and "...At most, the website will include a summary of the results."
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Blood Contamination in Fine Needle Biopsies for the Heparin Group
Description: H&E slides from passes 1, 2, and 3 will be reviewed. The amount of blood present on each H&E slide will be quantified by using image processing software (blood contamination area between passes).
Time Frame: Day 1 (biopsy tissue obtained)
Population: as for outcome 1
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Blood Contamination in Successive Fine Needle Biopsies Saline Group
Description: H&E slides from the pass 1, 2, and 3 will be reviewed. The amount of blood present on each H&E slide will be quantified by using image processing software (blood contamination area between passes).
Time Frame: Day 1 (biopsy tissue obtained)
Population: as for outcome 1
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Cellularity Captured in Successive Fine Needle Biopsies Saline Group
Description: H&E slides from the passes 1, 2, and 3 will be reviewed. The number of cells present on each H&E slide will be quantified by using image processing software.
  The data for this outcome will be calculated and reported as total number of cells divided by total area of the biopsy.
Time Frame: Day 1 (biopsy tissue obtained)
Population: as for outcome 1
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Participants Who Needed Repeated Endoscopic Ultrasound (EUS) Biopsy
Description: This outcome will report the number of participants who required a second EUS biopsy. Data was collected from health records.
Time Frame: 4 weeks (after initial biopsy)
Population: as for outcome 1
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

6. Other Pre Specified Outcome: Tissue Diagnosis
Description: H&E slides from the pass 1, 2, and 3 will be reviewed to see if a diagnosis can be made.
Time Frame: Day 1 (biopsy tissue obtained)
Population: as for outcome 1
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: No data is presented here because, with only 1 participant per arm, it is impossible to share this data, as doing so would conflict with the required informed consent language for ACTs, which says, "This website [ClinicalTrials.gov] will not include information that can identify you" and "...At most, the website will include a summary of the results."
Arm/Group | Heparin Priming Biopsies | Standard of Care (Saline)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-15): https://cdn.clinicaltrials.gov/large-docs/96/NCT04764396/Prot_SAP_000.pdf